CLINICAL TRIAL: NCT06170957
Title: The Effect of Modified Teat on Pain, Physiological Variables, and Stress Level During Heel Blood Collection in Mechanically Ventilated Term Newborns
Brief Title: Pacifier Use in Mechanically Ventilated Term Newborns
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hitit University (Other)
Responsible Party: Principal Investigator, Selen Ozakar Akca, Associate Professor Dr., Hitit University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HİTİTU
Record Dates: First submitted 2023-09-02; First posted 2023-12-14 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Pacifier
Keywords: newborn; mechanical ventilator; pacifier; physiological variables; pain; stress; cortisol level; invasive procedure (heel blood)
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Study
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): For the experimental group; A modified pacifier will be given to the newborn during the heel blood collection procedure.
  Interventions: Other: Modified pacifier
- Control group (No Intervention): For the control group; The newborn will not be given a modified pacifier during the heel blood collection procedure.

INTERVENTIONS:
Other: Modified pacifier — In this project, a pacifier produced from a modified pacifier shield made of polypropylene (PP), a biocompatible polymer, which is made suitable for intubation tube in newborns connected to mechanical ventilator, will be used in the light of literature information. No study on the modification of the pacifier shield has been found in the literature, and a utility model application (file number 2020/03477 dated 06 March 2020) was made for this pacifier shield, which is planned to be modified, and the utility model application was accepted on 04.02.2022.
  In the application of heel blood collection to newborns, a) before the procedure (20 minutes before), b) immediately before the procedure (20. minutes), c) during the procedure (between the 20th and 40th minutes), and d) 20 minutes after the procedure (40 minutes) will be evaluated once for each application, a total of four times.
  Arms: Experimental group

SUMMARY:
Newborns on mechanical ventilator; It is stated that they need to calm and soothe themselves, their coordination in sucking and swallowing reflexes is not good, they have aspiration risks, their weight gain and discharge are prolonged, and physiological stability is impaired. It is suggested that pacifiers can be used to reduce stress levels in these newborns. It has been observed that sterile gloves are used as pacifiers because the pacifier shields available in the market are not suitable for the intubation tube to calm the babies in the NICU. In order to reduce the stress level in newborns, developed in the light of this information, pacifier shields ergonomically suitable for intubation tube are designed. In this context, a modified pacifier shield was produced using a 3D printer from polypropylene (PP), a biocompatible polymer. It is aimed to examine the effects of using a modified pacifier on pain, physiological variables and stress level during heel blood collection in newborns who are connected to mechanical ventilator due to respiratory distress, considering that it would be more beneficial for newborns to adapt and use a model closest to the pacifier they will use in the future with the use of this modified pacifier.

DETAILED DESCRIPTION:
The neonatal period is defined as the first 28-day period of postnatal life. This period is stated as the transition period in which the newborn tries to adapt to extrauterine life, is sensitive and dynamic. One of the most common problems that occur during this period when the newborn experiences biochemical and physiological changes is respiratory failure. Respiratory failure is a cause of mortality and morbidity in the newborn. Therefore, the etiology should be determined quickly and intervened early. Newborns with or without respiratory failure need mechanical ventilation support to provide ventilation.

Mechanical ventilation is a life support system developed to support or fulfill normal lung functions. Mechanical ventilation is frequently used in infants hospitalized in the Neonatal Intensive Care Unit (NICU), to improve respiratory failure, to ensure adequate gas exchange, and to solve other problems. Newborns connected to mechanical ventilator, separation from the family in the intensive care environment, noise of the devices, invasive interventions, etc. They experience stress because they are exposed to painful stimuli due to many medical diagnosis and treatment procedures. These painful stimuli are a powerful source of stress. Stress is a factor that increases the susceptibility to physical and mental tension and illness due to physical, chemical or emotional factors. As a result of the stress experienced by newborns in the NICU due to painful stimuli, the secretion of glucocorticoids, especially cortisol, increases, long-term neurodevelopmental problems occur, and adverse events such as increase in heart rate, increase in catabolization and decrease in oxygen saturation values may occur.

Pain affects the endocrine system physiologically and activates the hypothalamic-pituitary-adrenal (HPA) axis, which is the body's main stress control mechanism. The function of the HPA axis and the resulting changes in cortisol levels in acute or chronic pain have been demonstrated by many studies. It has been reported that newborns with pain have higher cortisol levels and higher cortisol responses. It has been stated that this situation is associated with stressful events, there is an interaction between stress and pain, pain sensitivity increases in stressful situations, and the HPA axis is activated in case of stress, causing the release of glucocorticoids such as cortisol. In stressful situations, cortisol levels increase in newborns. Since the salivary cortisol level in newborns reflects the plasma cortisol level, it has been stated that determining the cortisol level is a reliable method in evaluating stress.

It is recommended to use pharmacological and non-pharmacological methods together to reduce pain and stress and minimize pain during short-term, mild and moderately painful procedures in newborns in the intensive care unit. Among non-pharmacological methods, non-nutritive sucking has vital importance in controlling pain, providing comfort and neurobehavioral control, increasing physiological stability and oxygenation, reducing stress, effective functioning of the digestive system and reducing the risk of aspiration. In the literature many painful procedures (circumcision, vaccination, IV catheterization, lumbar puncture test) of pacifier use It is reported that it provides an analgesic effect and reduces stress during In this context, it is stated that pacifier use has a calming effect and reduces stress for newborns and it is emphasized that it reduces salivary cortisol levels.

The endogenous analgesic effect of the pacifier; When a pacifier is placed in the mouth of the newborn, the sucking reflex is activated via a non-opioid mechanism, resulting in tactile sensitivity and stimulation of mechanical receptors. Since sucking prevents swallowing, it protects the baby against aspiration. Pacifier use in stressed newborns who also have tachycardia; It contributes to the calming of the newborn by causing stability in heart rate and increasing oxygenation. In this respect, the behavioral organization of newborns using pacifiers such as self-consolation and soothing develops, the time spent for sleep and wakefulness levels increase, the baby's energy consumption decreases and the discharge time is shortened. Smith et al. (2022) reviewed the NICU environment and published clinical practice guidelines recommending non-pharmacological methods to prevent pain and stress in neonates. Various non-pharmacological methods, including non-nutritive absorption, have been proposed in this guideline. The use of pacifiers in NICUs is recommended in the treatment plan of stressed newborns with poor sucking, swallowing and breathing coordination, as it helps neurobehavioral organization and maturation and supports calming. In addition to the benefits of pacifier use, there are also some risks such as otitis media, dental malocclusion, suffocation, allergies, increased caries risk, infections. However, when the mother and baby are separated and the benefits of the pacifier are evaluated, pacifier use is recommended for newborns. It is stated that the baby admitted to the NICU has a risk of losing its sucking reflexes as a result of being separated from the mother for a long time, and it is reported that non-nutritive sucking should be used to protect the sucking reflex, increase physiological stability and reduce stress. The Baby-Friendly Hospital Initiative, launched in 1990 by the World Health Organization (WHO) and the United Nations International Children's Emergency Fund (UNICEF) to promote and support breastfeeding, established the principles of "Ten Steps to Successful Breastfeeding". It was realized that these principles, which rejected the use of pacifiers in the future, did not take into account the separation of the mother and the baby, and it was suggested that this situation should be brought to the agenda. As a matter of fact, the "Ten Steps to Successful Breastfeeding" application was revised in 2013, and the use of pacifiers was recommended considering the special situations in which the newborn and mother were separated. In the literature prevent delays in nutritional development of newborns in ICUs who have to be separated from their mother, motor organization, supporting the development of neurobehavioral maturity levels, etc. The use of pacifiers is strongly recommended in justified cases. Painful and invasive procedures for follow-up, diagnostic and therapeutic purposes are an inevitable part of care in the intensive care unit. An effective pain and stress management is the main goal of nursing care and is based on a comprehensive assessment of the pain and stress of the newborn. Appropriate assessment of pain response and stress level directly affects and guides treatment. Physiological changes such as an increase in heart rate, respiratory rate, blood pressure and intracranial pressure, decrease in oxygen saturation, sweating in the palms, change in respiratory pattern, differentiation in skin color and pupil size are observed in newborns as a result of painful stimuli activating the sympathetic nervous system. The salivary cortisol level is a simple method used and recommended to evaluate the stress level of newborns. It is important to implement planned interventions in case of newborn stress. Nurses and other healthcare professionals have the responsibility to prevent or minimize the pain and stress of the newborn during procedures. The nurse's being with the patient for a long time contributes to the healing process by providing the evaluation and reduction of the patient's pain and stress.

Many studies have been found in the literature on the evaluation of pain and stress in newborns connected to mechanical ventilation, but it has been observed that there are no studies on the use of pacifiers in newborns connected to mechanical ventilation. Since pacifiers produced in the market are not suitable for mechanical ventilators it is planned to use the prototype of the pacifier shield designed by the researcher for newborn babies in this project.

ELIGIBILITY:
Inclusion Criteria:

* Newborns at 37-42 weeks who are connected to mechanical ventilator (intubated),
* Newborns on mechanical ventilator due to respiratory distress, Orotracheally connected to a mechanical ventilator,
* Intubated,
* Intubation tube without cuff, in the range of 3.5-4 mm diameter (in the calculation of intubation tube diameter in newborns, the calculation will be based on weight).
* Mechanical ventilator mode with "Pressure control/ Pressure control- Synchronized intermittent mandatory ventilation/ Synchronized intermittent mandatory ventilation" (PC-SIMV). There are also.)
* No neurological disorder,
* The babies of the families who agreed to participate in the study will be formed.

Exclusion Criteria:

* With neuromuscular disease,
* Structural and congenital malformations of the respiratory tract,
* İn the CPAP mask,
* Fed with orogastric,
* The intubation tube is fixed in the middle of the newborn, not the rim.
* Mechanical ventilator settings change frequently,
* Taking neuromuscular blocking drugs,
* Receiving high-dose inotropic support (Dopamine and/or Dobutamine 10mcg/kg/hour),
* Receiving medical treatment for chronic pain,

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Face, Legs, Activity, Cry, Consolability Pain Rating Scale | 40 minutes
  Pain level, min= 0 point, max= 10 point, 0 points = baby is calm and pain-free Score between 1-3 = baby has mild pain Score between 4-6 = the baby has moderate pain Score between 7-10 = the baby has serious pain
Physiological Variables | 40 minutes
  systolic-diastolic blood pressure (mmHg)
Physiological Variables | 40 minutes
  peak heart rate (min)
Physiological Variables | 40 minutes
  respiratory rate (min)
Physiological Variables | 40 minutes
  oxygen saturation value (%SpO2)
Measurement of Saliva Cortisol Level in Stress Assessment | 40 minutes
  Saliva level

IPD SHARING:
Plan to Share IPD: No
I Don't Plan to Share IPD

REFERENCES:
- [Background] Ancora G, Lago P, Garetti E, Merazzi D, Savant Levet P, Bellieni CV, Pieragostini L, Pirelli A. Evidence-based clinical guidelines on analgesia and sedation in newborn infants undergoing assisted ventilation and endotracheal intubation. Acta Paediatr. 2019 Feb;108(2):208-217. doi: 10.1111/apa.14606. Epub 2018 Dec 6. PMID 30290021
- [Background] Başara, S. G., Küçük, S. Mekanik ventilasyon tedavisi alan yenidoğanların bakımında hemşire: eğitim ve bilgi düzeyi ilişkisi. Acıbadem Üniversitesi Sağlık Bilimleri Dergisi. 2020; 11(2):330-336.
- [Background] Brummelte S, Grunau RE, Chau V, Poskitt KJ, Brant R, Vinall J, Gover A, Synnes AR, Miller SP. Procedural pain and brain development in premature newborns. Ann Neurol. 2012 Mar;71(3):385-96. doi: 10.1002/ana.22267. Epub 2012 Feb 28. PMID 22374882
- [Background] Cabral DM, Antonini SR, Custodio RJ, Martinelli CE Jr, da Silva CA. Measurement of salivary cortisol as a marker of stress in newborns in a neonatal intensive care unit. Horm Res Paediatr. 2013;79(6):373-8. doi: 10.1159/000351942. Epub 2013 Jun 20. PMID 23796826
- [Background] Çalışır, H., Güler, F. Yenidoğan yoğun bakım ünitesinde mekanik ventilasyon uygulanan prematüre bebeklere pozisyon verme. Türkiye Klinikleri Hemşirelik Bilimleri Dergisi. 2017; 9(3):227-232.
- [Background] Candia MF, Osaku EF, Leite MA, Toccolini B, Costa NL, Teixeira SN, Costa CR, Piana PA, Cristovam MA, Osaku NO. Influence of prone positioning on premature newborn infant stress assessed by means of salivary cortisol measurement: pilot study. Rev Bras Ter Intensiva. 2014 Apr-Jun;26(2):169-75. doi: 10.5935/0103-507x.20140025. PMID 25028952
- [Background] Cignacco E, Hamers JP, Stoffel L, van Lingen RA, Gessler P, McDougall J, Nelle M. The efficacy of non-pharmacological interventions in the management of procedural pain in preterm and term neonates. A systematic literature review. Eur J Pain. 2007 Feb;11(2):139-52. doi: 10.1016/j.ejpain.2006.02.010. Epub 2006 Apr 3. PMID 16580851
- [Background] Cingoz, İ. D., Ozyoruk, Ş., Husemoglu, B., Sahin, M. C.Surgery Dissector: Surgical Device Production With 3D Print Technology. Journal of Medical Innovation and Technology. 2019; 1(1):5-8.
- [Background] Cong X, Wu J, Vittner D, Xu W, Hussain N, Galvin S, Fitzsimons M, McGrath JM, Henderson WA. The impact of cumulative pain/stress on neurobehavioral development of preterm infants in the NICU. Early Hum Dev. 2017 May;108:9-16. doi: 10.1016/j.earlhumdev.2017.03.003. Epub 2017 Mar 23. PMID 28343092
- [Background] Coviello C, Popple Martinez M, Drovandi L, Corsini I, Leonardi V, Lunardi C, Antonelli C, Pratesi S, Dani C. Painful procedures can affect post-natal growth and neurodevelopment in preterm infants. Acta Paediatr. 2018 May;107(5):784-790. doi: 10.1111/apa.14222. Epub 2018 Feb 6. PMID 29341252
- [Background] Crellin D, Harrison D, Santamaria N, Babl FE. Comparison of the Psychometric Properties of the FLACC Scale, the MBPS and the Observer Applied Visual Analogue Scale Used to Assess Procedural Pain. J Pain Res. 2021 Mar 31;14:881-892. doi: 10.2147/JPR.S267839. eCollection 2021. PMID 33833566
- [Background] Duman, N. Prematürede solunum problemleri ve yönetimi. Klinik Tıp Pediatri Dergisi. 2017;9(4):17-32.
- [Background] Foster JP, Psaila K, Patterson T. Non-nutritive sucking for increasing physiologic stability and nutrition in preterm infants. Cochrane Database Syst Rev. 2016 Oct 4;10(10):CD001071. doi: 10.1002/14651858.CD001071.pub3. PMID 27699765
- [Background] Eroğlu, A., Arslan, S. Yenidoğanda ağrının algılanması, değerlendirilmesi ve yönetimi. Düzce Üniversitesi Sağlık Bilimleri Enstitüsü Dergisi. 2018; 8(1):52-60.
- [Background] Garcia-Rodriguez MT, Bujan-Bravo S, Seijo-Bestilleiro R, Gonzalez-Martin C. Pain assessment and management in the newborn: A systematized review. World J Clin Cases. 2021 Jul 26;9(21):5921-5931. doi: 10.12998/wjcc.v9.i21.5921. PMID 34368310
- [Background] Gederi A, Coomaraswamy K, Turner PJ. Pacifiers: a review of risks vs benefits. Dent Update. 2013 Mar;40(2):92-4, 97-8, 101. doi: 10.12968/denu.2013.40.2.92. PMID 23600033
- [Background] Tekgunduz KS, Polat S, Gurol A, Apay SE. Oral Glucose and Listening to Lullaby to Decrease Pain in Preterm Infants Supported with NCPAP: A Randomized Controlled Trial. Pain Manag Nurs. 2019 Feb;20(1):54-61. doi: 10.1016/j.pmn.2018.04.008. Epub 2018 Dec 13. PMID 29776872
- [Background] Harding, C. M., Law, J., Pring, T. The use of non-nutritive sucking to promote functional sucking skills in premature infants: an exploratory trial. Infant. 2006;2(6):238-240.
- [Background] Hellhammer DH, Wust S, Kudielka BM. Salivary cortisol as a biomarker in stress research. Psychoneuroendocrinology. 2009 Feb;34(2):163-171. doi: 10.1016/j.psyneuen.2008.10.026. Epub 2008 Dec 18. PMID 19095358
- [Background] Janevski MR, Vujicic AD, Dukic SM. Salivary Cortisol as a Biomarker of Stress in Mothers and their Low Birth Weight Infants and Sample Collecting Challenges. J Med Biochem. 2016 Apr;35(2):118-122. doi: 10.1515/jomb-2015-0015. Epub 2016 May 9. PMID 28356870
- [Background] Jenik AG, Vain N. The pacifier debate. Early Hum Dev. 2009 Oct;85(10 Suppl):S89-91. doi: 10.1016/j.earlhumdev.2009.08.025. Epub 2009 Sep 17. PMID 19762175
- [Background] Krishnan L. Pain relief in neonates. J Neonatal Surg. 2013 Apr 1;2(2):19. eCollection 2013 Apr-Jun. No abstract available. PMID 26023439
- [Background] Lee, J., Lee, H., Cheon, K. H., Park, C., Jang, T. S., Kim, H. E., Jung, H. D.Fabrication of poly (lactic acid)/Ti composite scaffolds with enhanced mechanical properties and biocompatibility via fused filament fabrication (FFF)-based 3D printing. Additive Manufacturing. 2019; 30:100883.
- [Background] Lee K, Oh H, Suh Y, Seo W. Patterns and clinical correlates of pain among brain injury patients in critical care assessed with the critical care pain observation tool. Pain Manag Nurs. 2013 Dec;14(4):259-267. doi: 10.1016/j.pmn.2011.05.005. Epub 2011 Jul 20. PMID 24315249
- [Background] Lubbe W, Ten Ham-Baloyi W. When is the use of pacifiers justifiable in the baby-friendly hospital initiative context? A clinician's guide. BMC Pregnancy Childbirth. 2017 Apr 27;17(1):130. doi: 10.1186/s12884-017-1306-8. PMID 28449646
- [Background] Maas C, Ringwald C, Weber K, Engel C, Poets CF, Binder G, Bassler D. Relationship of salivary and plasma cortisol levels in preterm infants: results of a prospective observational study and systematic review of the literature. Neonatology. 2014;105(4):312-8. doi: 10.1159/000357555. Epub 2014 Mar 5. PMID 24603497
- [Background] McCarthy AM, Kleiber C, Hanrahan K, Zimmerman MB, Westhus N, Allen S. Factors explaining children's responses to intravenous needle insertions. Nurs Res. 2010 Nov-Dec;59(6):407-16. doi: 10.1097/NNR.0b013e3181f80ed5. PMID 20962698
- [Background] McLean MA, Nakajima L, Chau CMY, Weinberg J, Synnes AR, Miller SP, Grunau RE. Cortisol levels are related to neonatal pain exposure in children born very preterm at age 18 months in two independent cohorts. Paediatr Neonatal Pain. 2023 May 29;5(3):86-95. doi: 10.1002/pne2.12112. eCollection 2023 Sep. PMID 37744280
- [Background] Mitsuishi, H., Okamura, H., Moriguchi, Y., Aoki, Y. The validity of the salivary cortisol analysis method using the cube reader in japanese university students. Japanese Psychological Research. 2022; 1-10.
- [Background] Morelius E, He HG, Shorey S. Salivary Cortisol Reactivity in Preterm Infants in Neonatal Intensive Care: An Integrative Review. Int J Environ Res Public Health. 2016 Mar 18;13(3):337. doi: 10.3390/ijerph13030337. PMID 26999185
- [Background] Morelius E, Theodorsson E, Nelson N. Stress at three-month immunization: parents' and infants' salivary cortisol response in relation to the use of pacifier and oral glucose. Eur J Pain. 2009 Feb;13(2):202-8. doi: 10.1016/j.ejpain.2008.03.016. Epub 2008 May 16. PMID 18486508
- [Background] Nees F, Loffler M, Usai K, Flor H. Hypothalamic-pituitary-adrenal axis feedback sensitivity in different states of back pain. Psychoneuroendocrinology. 2019 Mar;101:60-66. doi: 10.1016/j.psyneuen.2018.10.026. Epub 2018 Oct 26. PMID 30414593
- [Background] Neiva FC, Leone CR, Leone C, Siqueira LL, Uema KA, Evangelista D, Delgado S, Rocha A, Buhler KB. Non-nutritive sucking evaluation in preterm newborns and the start of oral feeding: a multicenter study. Clinics (Sao Paulo). 2014 Jun;69(6):393-7. doi: 10.6061/clinics/2014(06)05. PMID 24964303
- [Background] Nyqvist KH, Haggkvist AP, Hansen MN, Kylberg E, Frandsen AL, Maastrup R, Ezeonodo A, Hannula L, Haiek LN; Baby-Friendly Hospital Initiative Expert Group. Expansion of the baby-friendly hospital initiative ten steps to successful breastfeeding into neonatal intensive care: expert group recommendations. J Hum Lact. 2013 Aug;29(3):300-9. doi: 10.1177/0890334413489775. Epub 2013 May 31. PMID 23727630
- [Background] Ojha S, Abramson J, Dorling J. Sedation and analgesia from prolonged pain and stress during mechanical ventilation in preterm infants: is dexmedetomidine an alternative to current practice? BMJ Paediatr Open. 2022 May;6(1):e001460. doi: 10.1136/bmjpo-2022-001460. PMID 36053596
- [Background] Pinelli, J., Symington, A. Non-nutritive sucking for promoting physiologic stability and nutrition in preterm infants. Evidence-based Child Health: A Cochrane Review Journal, 2011;6(4):1134-1169.
- [Background] Popowicz H, Kwiecien-Jagus K, Olszewska J, Medrzycka-Dabrowska WA. Pain Scales in Neonates Receiving Mechanical Ventilation in Neonatal Intensive Care Units - Systematic Review. J Pain Res. 2020 Jul 24;13:1883-1897. doi: 10.2147/JPR.S248042. eCollection 2020. PMID 32801846
- [Background] Popowicz H, Medrzycka-Dabrowska W, Kwiecien-Jagus K, Kamedulska A. Knowledge and Practices in Neonatal Pain Management of Nurses Employed in Hospitals with Different Levels of Referral-Multicenter Study. Healthcare (Basel). 2021 Jan 5;9(1):48. doi: 10.3390/healthcare9010048. PMID 33466529
- [Background] Poyak J. Effects of pacifiers on early oral development. Int J Orthod Milwaukee. 2006 Winter;17(4):13-6. PMID 17256438
- [Background] Provenzi L, Giusti L, Fumagalli M, Tasca H, Ciceri F, Menozzi G, Mosca F, Morandi F, Borgatti R, Montirosso R. Pain-related stress in the Neonatal Intensive Care Unit and salivary cortisol reactivity to socio-emotional stress in 3-month-old very preterm infants. Psychoneuroendocrinology. 2016 Oct;72:161-5. doi: 10.1016/j.psyneuen.2016.07.010. Epub 2016 Jul 10. PMID 27428089
- [Background] Ramos, M. C. M., de Candido, L. K., Costa, T., Leite, A. C., Manzo, B. F., Duarte, E. D., Harrison, D., Bueno, M. Painful procedures and analgesia in hospitalized newborns: A prospective longitudinal study. Journal of Neonatal Nursing. 2019;25(1):26-31.
- [Background] Redmann AJ, Wang Y, Furstein J, Myer CM 3rd, de Alarcon A. The use of the FLACC pain scale in pediatric patients undergoing adenotonsillectomy. Int J Pediatr Otorhinolaryngol. 2017 Jan;92:115-118. doi: 10.1016/j.ijporl.2016.11.016. Epub 2016 Nov 24. PMID 28012511
- [Background] Rocha CR, Verga KE, Sipsma HL, Larson IA, Phillipi CA, Kair LR. Pacifier Use and Breastfeeding: A Qualitative Study of Postpartum Mothers. Breastfeed Med. 2020 Jan;15(1):24-28. doi: 10.1089/bfm.2019.0174. Epub 2019 Dec 20. PMID 31859530
- [Background] Rocha VA, Silva IA, da Silveira Cruz-Machado S, Bueno M. Painful procedures and pain management in newborns admitted to an intensive care unit. Rev Esc Enferm USP. 2021 Oct 29;55:e20210232. doi: 10.1590/1980-220X-REEUSP-2021-0232. eCollection 2021. English, Portuguese. PMID 34714319
- [Background] Senayli, Y., Ozkan, F., Şenaylı, A., Bicakci, U. Evaluation of postoperative pain in children with FLACC pain scale in Turkish translation. Turkiye Klinikleri Journal of Anesthesiology Reanimation. 2006;4(1):1-4.
- [Background] Sılay, F., Akyol, A. Yoğun bakım ünitelerinde sedasyon-ajitasyon ve ağrı değerlendirmesinde kullanılan iki ölçüm aracının türkçe'ye uyarlanması: geçerlilik ve güvenilirlik çalışması. Yoğun Bakım Hemşireliği Dergisi. 2018;22(2):50-65.
- [Background] Sixtus RP, Gray C, Berry MJ, Dyson RM. Preterm-born individuals: a vulnerable population at risk of cardiovascular morbidity and mortality during thermal extremes? Exp Physiol. 2023 Aug;108(8):1011-1025. doi: 10.1113/EP091152. Epub 2023 Apr 21. PMID 37084061
- [Background] Smallwood CD, Davis MD. Year in Review 2018: Pediatric Mechanical Ventilation. Respir Care. 2019 Jul;64(7):855-863. doi: 10.4187/respcare.07029. PMID 31243160
- [Background] Smith HAB, Besunder JB, Betters KA, Johnson PN, Srinivasan V, Stormorken A, Farrington E, Golianu B, Godshall AJ, Acinelli L, Almgren C, Bailey CH, Boyd JM, Cisco MJ, Damian M, deAlmeida ML, Fehr J, Fenton KE, Gilliland F, Grant MJC, Howell J, Ruggles CA, Simone S, Su F, Sullivan JE, Tegtmeyer K, Traube C, Williams S, Berkenbosch JW. 2022 Society of Critical Care Medicine Clinical Practice Guidelines on Prevention and Management of Pain, Agitation, Neuromuscular Blockade, and Delirium in Critically Ill Pediatric Patients With Consideration of the ICU Environment and Early Mobility. Pediatr Crit Care Med. 2022 Feb 1;23(2):e74-e110. doi: 10.1097/PCC.0000000000002873. PMID 35119438
- [Background] Sönmez Düzkaya, D. Pediatrik yoğun bakımda ventilatör ilişkili pnömoninin önlenmesinde hemşirenin rolü. The Journal of Pediatric Research.2014;1(2):54-61.
- [Background] Tennant F. The physiologic effects of pain on the endocrine system. Pain Ther. 2013 Dec;2(2):75-86. doi: 10.1007/s40122-013-0015-x. Epub 2013 Aug 20. PMID 25135146
- [Background] Timmers I, Kaas AL, Quaedflieg CWEM, Biggs EE, Smeets T, de Jong JR. Fear of pain and cortisol reactivity predict the strength of stress-induced hypoalgesia. Eur J Pain. 2018 Aug;22(7):1291-1303. doi: 10.1002/ejp.1217. Epub 2018 Apr 19. PMID 29577522
- [Background] Turan, T., Erdoğan, Ç. Yenidoğan Yoğun Bakım Ünitesindeki Prematüre Bebeğin Gelişiminin Desteklenmesi.Hemşirelik Akademik Araştırma Dergisi. 2018;4(2):127-132.
- [Background] Valeri BO, Holsti L, Linhares MB. Neonatal pain and developmental outcomes in children born preterm: a systematic review. Clin J Pain. 2015 Apr;31(4):355-62. doi: 10.1097/AJP.0000000000000114. PMID 24866853
- [Background] Venkatesh B, Cohen J, Hickman I, Nisbet J, Thomas P, Ward G, Hall J, Prins J. Evidence of altered cortisol metabolism in critically ill patients: a prospective study. Intensive Care Med. 2007 Oct;33(10):1746-53. doi: 10.1007/s00134-007-0727-7. Epub 2007 Jun 9. PMID 17558491
- [Background] Verweij LM, Kivits JTS, Weber F. The performance of the heart rate variability-derived Newborn Infant Parasympathetic Evaluation Index as a measure of early postoperative pain and discomfort in infants-A prospective observational study. Paediatr Anaesth. 2021 Jul;31(7):787-793. doi: 10.1111/pan.14188. Epub 2021 May 6. PMID 33811710
- [Background] Vu-Ngoc H, Uyen NCM, Thinh OP, Don LD, Danh NVT, Truc NTT, Vi VT, Vuong NL, Huy NT, Duong PDT. Analgesic effect of non-nutritive sucking in term neonates: A randomized controlled trial. Pediatr Neonatol. 2020 Feb;61(1):106-113. doi: 10.1016/j.pedneo.2019.07.003. Epub 2019 Aug 8. PMID 31474462
- [Background] Watanabe E, Kuchta K, Kimura M, Rauwald HW, Kamei T, Imanishi J. Effects of bergamot ( Citrus bergamia (Risso) Wright & Arn.) essential oil aromatherapy on mood states, parasympathetic nervous system activity, and salivary cortisol levels in 41 healthy females. Forsch Komplementmed. 2015;22(1):43-9. doi: 10.1159/000380989. Epub 2015 Feb 19. PMID 25824404
- [Background] Wu HP, Yang L, Lan HY, Peng HF, Chang YC, Jeng MJ, Liaw JJ. Effects of Combined Use of Mother's Breast Milk, Heartbeat Sounds, and Non-Nutritive Sucking on Preterm Infants' Behavioral Stress During Venipuncture: A Randomized Controlled Trial. J Nurs Scholarsh. 2020 Sep;52(5):467-475. doi: 10.1111/jnu.12571. Epub 2020 Jun 20. PMID 32564489